CLINICAL TRIAL: NCT04703764
Title: A Dose Blocked-randomized, Double Blind, Placebo-controlled, Multiple Dosing, Phase I Clinical Trial to Evaluate the Safety and Pharmacokinetic/Pharmacodynamic Characteristics of HSG4112 After Oral Administration in Healthy and Obese Adult Subjects
Brief Title: A Study to Investigate the Safety and Pharmacokinetic/Pharmacodynamic Characteristics of HSG4112
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Glaceum (Industry)
Collaborators: Kyungpook National University Hospital (Other); Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSG4112-P1-03
Record Dates: First submitted 2020-12-16; First posted 2021-01-11 (Actual); Last update posted 2022-09-09 (Actual); Status verified 2022-09

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HSG4112 480 mg (Experimental): 60 mg HSG4112 tablet, 8 tablets, once-daily, 14-day multiple oral administration
  Interventions: Drug: HSG4112
- Placebo 480 mg (Placebo Comparator): 60 mg placebo tablet, 8 tablets, once-daily, 14-day multiple oral administration
  Interventions: Drug: Placebo
- HSG4112 720 mg (Experimental): 60 mg HSG4112 tablet, 12 tablets, once-daily, 14-day multiple oral administration
  Interventions: Drug: HSG4112
- Placebo 720 mg (Placebo Comparator): 60 mg placebo tablet, 12 tablets, once-daily, 14-day multiple oral administration
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HSG4112 — Once-daily, 14-day multiple oral administration
  Other Names: 2-(8,8 dimethyl 2,3,4,8,9,10 hexahydropyrano[2,3 f]chromen 3 yl) 5 ethoxyphenol
  Arms: HSG4112 480 mg; HSG4112 720 mg
Drug: Placebo — Once-daily, 14-day multiple oral administration
  Arms: Placebo 480 mg; Placebo 720 mg

SUMMARY:
1. Study Objective

   <Part 1> To evaluate the safety and pharmacokinetic/pharmacodynamic characteristics of HSG4112 after multiple oral administration in healthy female subjects.

   <Part 2> To evaluate the safety and pharmacokinetic/pharmacodynamic characteristics of HSG4112 after multiple oral administration in obese subjects.
2. Background

   The previous phase 1 clinical trials investigating HSG4112 only included healthy male subjects, and food effect was observed in theses studies - the plasma exposure to HSG4112 following administration under fed conditions was approximately 2.5 times higher compared to the exposure following administration under fasted conditions. Therefore, this study is designed to evaluate the safety of HSG4112 in healthy female subjects and obese subjects following the administration of HSG4112 under fed conditions.
3. Study Design and Plan

<Part 1> This study is a dose block-randomized, double-blind, placebo-controlled, multiple dosing, phase 1 clinical study. A unique randomization number will be assigned to each subject deemed eligible to participate in the study based on the inclusion/exclusion criteria. Each subject will be randomized to one of the two dose groups. In each dose group, 8 subjects will be randomized to receive HSG4112 and 2 subjects will be randomized to receive placebo. The subjects will be studied in a double-blind manner and will receive the investigational product (i.e., HSG4112 or placebo) via once-daily oral administration for 14 consecutive days. After the Post-Study Visit of the last volunteer in the 480 mg dose group, the Investigator will review all the available safety data in a blinded manner to ensure if it is safe to proceed with the 720 mg dose group. In order to evaluate safety and tolerability, assessments, such as vital signs, 12-lead ECG, laboratory test, pregnancy test, physical examination, and adverse event monitoring will be performed. Blood samples will be collected to evaluate the pharcokinetic/pharmacodynamic characteristics of HSG4112.

<Part 2> This study is a dose block-randomized, double-blind, placebo-controlled, multiple dosing, phase 1 clinical study. A unique randomization number will be assigned to each subject deemed eligible to participate in the study based on the inclusion/exclusion criteria. Each subject will be randomized to one of the two dose groups. In each dose group, 8 subjects will be randomized to receive HSG4112 and 2 subjects will be randomized to receive placebo. The subjects will be studied in a double-blind manner and will receive the investigational product (i.e., HSG4112 or placebo) via once-daily oral administration for 14 consecutive days. In order to evaluate safety and tolerability, assessments, such as vital signs, 12-lead ECG, laboratory test, pregnancy test, physical examination, and adverse event monitoring will be performed. Blood samples will be collected to evaluate the pharcokinetic/pharmacodynamic characteristics of HSG4112.

ELIGIBILITY:
<Part 1>

Inclusion Criteria:

1. Able to comprehend and willing to sign an informed consent form approved by the IRB before screening.
2. Females between 19 and 50 years of age at screening.
3. Body mass index (BMI) between 18.0 and 24.9.

   * BMI (kg/m2) = Body weight (kg) / {Height (m)2}
4. In good health, determined by no clinically significant findings from medical history, physical examination, vital signs, 12-lead electrocardiogram, and clinical laboratory evaluations at screening, or subjects who are deemed acceptable by the Investigator regardless of the test results.
5. Not pregnant or lactating, with a regular menstrual cycle (i.e., 28±7 days).

Exclusion Criteria:

1. Significant history or clinical manifestation of any hepatic, kidney, neurological, immune, respiratory, endocrine, hematological, neoplastic, or cardiovascular disease, or psychiatric disorder (e.g., mood disorder, obsessive-compulsive disorder).
2. History of stomach or intestinal disorders (e.g., Chrons disease, ulcer) or surgeries - not including appendectomy, hemorrhoidectomy, or herniotomy - which may affect the pharmacokinetic or pharmacodynamic evaluation of the investigational product.
3. Significant history or clinical manifestation of hypersensitivity to any drug compound (e.g., licorice, aspirin, antibiotics).
4. One or more of the following laboratory test results at screening:

   * ALT > 60 IU/L
   * Glucose (fasting) > 100 mg/dL or < 70 mg/dL
5. Systolic blood pressure of < 90 mmHg or > 150 mmHg, or diastolic blood pressure of < 60 mgHg or > 100 mmHg as determined by vital signs monitored after resting in sitting position for at least 3 minutes.
6. History of drug/chemical abuse or tested positive in urine drug screen.
7. Use or intend to use any prescription medications/products or phytotherapeutic/herbal/plant-derived preparations within 14 days prior to dosing, or any nonprescription medications/products (i.e., over-the-counter (OTC) drugs), health products, or vitamins within 7 days prior to dosing, unless deemed acceptable by the Investigator.
8. Participation in any clinical study or bioequivalence study involving administration of an investigational drug, including any study investigating HSG4112, within 6 months prior to dosing (i.e., within 6 months of the last dose from the previous study).
9. Whole blood donation within 2 months prior to dosing, plasma/platelet donation within 1 month prior to dosing, or receipt of blood products within 1 month prior to dosing.
10. Smoker. However, participation is acceptable if the subject has quit smoking at least 3 months prior to dosing.
11. Alcohol consumption of > 21 units/week (1 unit = 10 g of pure alcohol) or unable to abstain from consuming alcohol during the study period.
12. Ingestion of grapefruit-containing foods or beverages 24 hours prior to dosing until discharge, or unable to abstain from ingesting such foods or beverages during the same period.
13. Unable to abstain from caffeine-containing foods or beverages (e.g., coffee, tea (e.g., black tea, green tea), soft drinks, coffee milk, energy drinks, sports drinks) during the admission period.
14. One or more of the following contraception- or pregnancy-related exclusion criteria:

    * Females of childbearing potential who are unable or unwilling to use acceptable contraceptive methods during the study period. 'A female of childbearing potential' refers to premenopausal females (i.e., females who who have experienced amenorrhoea for 12 months or longer) who are capable of becoming pregnant following menarche and have not been surgically sterilized (e.g., hysterectomy, bilateral tubal ligation, bilateral salpingectomy, bilateral oophorectomy).

      * Acceptable contraceptive methods include: intrauterine device that has been proven highly effective, physical contraception (e.g., diaphragm, uterine cap, condom) used with chemical sterilization (e.g., spermicide), or surgical sterilization (e.g., vasectomy, hysterectomy, tubal ligation, salpingectomy) of the subject or the subject's male partner.
    * Intend to use hormonal contraceptive methods during the study period.
    * Females of childbearing potential who have tested positive for pregnancy, determined by the pregnancy test.
15. Subjects who, in the opinion of the Investigator, should not participate in this study based on clinical laboratory test results or other reasons.

<Part 2>

Inclusion Criteria:

1. Able to comprehend and willing to sign an informed consent form approved by the IRB before screening.
2. Adults between 19 and 50 years of age at screening.
3. Body mass index (BMI) of 30.0 or higher, with a waist circumference of 90 cm or higher for males and 85 cm or higher for females.

   * BMI (kg/m2) = Body weight (kg) / {Height (m)2}
4. Deemed acceptable by the Investigator through medical history, physical examination, vital signs, 12-lead ECG, and clinical laboratory evaluations at screening, or subjects who are deemed acceptable by the Investigator regardless of the test results.

Exclusion Criteria:

1. Significant history or clinical manifestation of any hepatic, kidney, neurological, immune, respiratory, endocrine, hematological, neoplastic, cardiovascular, psychiatric diseases or compulsive disorder.
2. History of stomach or intestinal disorders (e.g., Chrons disease, ulcer) or surgeries - not including appendectomy, hemorrhoidectomy, or herniotomy - which may affect the pharmacokinetic or pharmacodynamic evaluation of the investigational product.
3. Significant history or clinical manifestation of hypersensitivity to any drug compound (e.g., licorice, aspirin, antibiotics).
4. One or more of the following laboratory test results at screening:

   * AST > 100 IU/L
   * ALT > 100 IU/L
   * Cholesterol > 300 mg/dL (subjects who need treatment for their cholesterol level will be excluded)
   * Triglyceride > 300 mg/dL
   * Glucose (fasting) of 126 mg/dL or higher
5. Systolic blood pressure of < 90 mmHg or > 150 mmHg, or diastolic blood pressure of < 60 mgHg or > 100 mmHg as determined by vital signs monitored after resting in sitting position for 3 minutes or longer.
6. History of drug/chemical abuse or tested positive in urine drug screen.
7. Use or intend to use any prescription medications/products or phytotherapeutic/herbal/plant-derived preparations 14 days prior to dosing, or any nonprescription medications/products (i.e., over-the-counter (OTC) drugs), health products, or vitamins 7 days prior to dosing, unless deemed acceptable by the Investigator.
8. Participation in any clinical study or bioequivalence study involving administration of an investigational drug, including any study investigating HSG4112, 6 months prior to dosing (i.e., within 6 months of the last dose from the previous study).
9. Whole blood donation within 2 months prior to dosing, plasma/platelet donation within 1 month prior to dosing, or receipt of blood products within 1 month prior to dosing.
10. Smoker. However, participation is acceptable if the subject has quit smoking 3 months prior to dosing.
11. Alcohol consumption of > 21 units/week (1 unit = 10 g of pure alcohol) or unable to abstain from consuming alcohol during the study period.
12. Ingestion of grapefruit-containing foods or beverages 24 hours prior to dosing until discharge, or unable to abstain from ingesting such foods or beverages during the same period.
13. Unable to abstain from caffeine-containing foods or beverages (e.g., coffee, tea (black tea, green tea, etc.), soft drinks, coffee milk, energy drinks, sports drinks) during the admission period.
14. Females who have tested positive in a urine HCG test, are pregnant, or lactating before the dosing of an investigational product, excluding females who have experienced amenorrhoea for 12 months or longer or have been surgically sterilized (e.g., hysterectomy, bilateral tubal ligation, bilateral salpingectomy, bilateral oophorectomy).
15. Unable or unwilling to use contraceptive methods during the study period, up to 30 days after the last day of dosing.

    * Acceptable contraceptive methods include:

      * Use of an intrauterine device that has been proven highly effective by the subject or the subject's partner.
      * Physical contraception (e.g., diaphragm, uterine cap, condom) used with chemical sterilization (e.g., spermicide)
      * Surgical sterilization of the subject or the subject's partner (e.g., vasectomy, hysterectomy, tubal ligation, salpingectomy).
16. Subjects who, in the opinion of the Investigator, should not participate in in this study based on clinical laboratory test results or other reasons.

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2022-01-20 (Actual); Study Completion 2022-02-03 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic Assessment by Area Under the Plasma Concentration-Time Curve of HSG4112 Over Dosing Interval | Hour 0 to 24
  Area under the plasma concentration-time curve of HSG4112 over dosing interval (AUCtau,ss)
Pharmacokinetic Assessment by Area Under the Plasma Concentration-Time Curve of HSG4112 from Time Zero to the Last Measurable Point | Hour 0 to 192
  Area under the plasma concentration-time curve from time zero to the last measurable point (AUClast)
Pharmacokinetic Assessment by Area Under the Plasma Concentration-Time Curve of HSG4112 from Time Zero to Infinity | Hour 0 to 192
  Area under the plasma concentration-time curve from time zero to infinity (AUCinf)
Pharmacokinetic Assessment by Maximum and Minimum Plasma Concentration of HSG4112 | Hour 0 to 192
  Maximum and minimum plasma concentration of HSG4112 (Cmax,ss; Cmin,ss)
Pharmacokinetic Assessment by Time to Maximum Observed Plasma Concentration of HSG4112 | Hour 0 to 192
  Time to maximum observed plasma concentration of HSG4112 (Tmax)
Pharmacokinetic Assessment by Half-Life of HSG4112 | Hour 0 to 192
  Half-life of HSG4112 (T1/2)
Pharmacokinetic Assessment by Oral Clearance of HSG4112 | Hour 0 to 192
  Oral clearance of HSG4112 (CLss/F)
Pharmacokinetic Assessment by Volume of Distribution of HSG4112 | Hour 0 to 192
  Volume of distribution of HSG4112 (Vd/F)
Safety and Tolerability Assessment by Number of Participants with Change in Vital Signs | Day 1, 14, and post-study visit
  Number of participants with clinically significant change in vital signs including blood pressure (mmHg) measured with blood pressure monitor, heart rate (beats per minute) measured with pulse oximeter, and body temperature (degrees Celcius) measured with thermometer
Safety and Tolerability Assessment by Number of Participants with Change in 12-Lead Electrocardiogram | Day -1, 11, and post-study visit
  Number of participants with clinically significant change in 12-lead electrocardiogram
Safety and Tolerability Assessment by Number of Participants with Change in Laboratory Test | Day -1, 8, 13, 15, 17, and post-study visit
  Number of participants with clinically significant change in laboratory test assessed through hematology, blood biochemistry, urinalysis, and blood coagulation test
Safety and Tolerability Assessment by Pregnancy Test | Day -1, 11, and post-study visit
  Monitoring the pregnancy status of participants through urine pregnancy test by measuring the level of human chorionic gonadotropin
Safety and Tolerability Assessment by Number of Patients with Change in Physical Examination | Day -1, 1 to 14, 17, and post-study visit
  Number of participants with clinically significant change in physical examination

SECONDARY OUTCOMES:
Pharmacodynamic Assessment by Change of Body Weight in Healthy Subjects | Day -1, 8, 15, and 22
  Assessment of the weight loss effect of HSG4112 by change of observed body weight compared to baseline (kg)
Pharmacodynamic Assessment by Change of Body Weight in Obese Subjects | Day 1 to 17, 18, 20, and 22
  Assessment of the weight loss effect of HSG4112 by change of observed body weight compared to baseline (kg)
Pharmacodynamic Assessment by Change of Waist Circumference | Day -1, 8, 15, and 22
  Assessment of the weight loss effect of HSG4112 by change of observed waist circumference compared to baseline (cm)
Pharmacodynamic Assessment by Change of Biomarkers | Day 1 and 14 pre-dose
  Assessment of the weight loss effect of HSG4112 by measurement of biomarkers including leptin, adiponectin, insulin, C-peptide (connecting peptide), IL6 (interleukin 6), TNF-alpha (tumor necrosis factor alpha), and CCL2 (C-C motif ligand 2) from baseline to day of last dosing
Pharmacodynamic Assessment by Change of Fat Mass and Body Fat Percentage | Day 1, 8, 15, and 22
  Assessment of the weight loss effect of HSG4112 by change of fat mass (kg) and body fat percentage (%) compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Young-Ran Yoon, Principal Investigator — Kyungpook National University Hospital
Locations (2):
- South Korea (2):
  - Kyungpook National University Hospital, Daegu
  - Seoul National University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No